CLINICAL TRIAL: NCT01806012
Title: Use of the Enseal Intrument for Laparoscopic Supracervical Hysterectomy: a Randomized, Single-Blinded Study Comparing the Efficacy to the Routine Procedure
Brief Title: Use of the Enseal Intrument for Laparoscopic Supracervical Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard Kraemer, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05022013
Record Dates: First submitted 2013-02-19; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Indications for Laparoscopic Supracervical Hysterectomy
Keywords: Supracervical Hysterectomy; Leiomyomas; Adenomyosis
MeSH Terms: conditions — Leiomyoma; Adenomyosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enseal (Experimental): Tissue sealing with Enseal device
  Interventions: Device: Sealing tissue with the Enseal device
- Supracervical hysterectomy using conventional instruments (Active Comparator): Supracervical hysterectomy using conventional instruments
  Interventions: Procedure: Conventional supracervical hysterectomy

INTERVENTIONS:
Device: Sealing tissue with the Enseal device
  Arms: Enseal
Procedure: Conventional supracervical hysterectomy
  Arms: Supracervical hysterectomy using conventional instruments

SUMMARY:
The use of the EnSeal® instrument for laparoscopic supracervical hysterectomy in a randomized, single-blinded comparison to the conventional procedure. The objective of the study is to investigate if the use of the Enseal sealing instrument for supracervical hysterectomy leads to a shortening of the operation time.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Indication for supracervical hysterectomy without additional surgical procedures (i. e. oophorectomy)
* Willingness and capability to comply with all study tests, procedures, and assessment tools
* Capability of providing informed consent.

Exclusion Criteria:

* History of, or evidence of, gynecologic malignancy within the past five years
* Pace maker, internal defibrilator/cardioconverter
* Impaired coagulation parameters
* Unwillingness to be randomized to treatment
* History of median laparotomy
* Intraabdominal adhesions
* Requirement for open laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Operation time | Day 1
  The following times were documented: total operation time; T1 = start of the operation until cornual structures were ready to be dissected; T2 = the time from the first coagulation and cutting of the cornual structures until the complete preparation of each parametrial side directly before cervical detachment; T3 = time needed for the cervical detachment and subsequent steps (morcellation, closure of trocar sites) until the end of the surgical procedure.

SECONDARY OUTCOMES:
Blood loss | Day 2
  The perioperative blood loss (ΔHb) was calculated using the comparison of the preoperative red blood cells (RBC) versus the RBC on the first post-operative day. The intraoperative blood loss was measured by the suction unit (categories: < 50 ml, 50 - 100 ml, > 100 ml) and by the number of applied blood transfusions.
Post-operative pain | Day 2
  Post-operative pain was documented according to a visual analog pain scale from 1 (no pain) to 10 (maximum pain) during hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- University Women' Clinic Tübingen, Tübingen, Germany

REFERENCES:
- [Derived] Rothmund R, Kraemer B, Brucker S, Taran FA, Wallwiener M, Zubke A, Wallwiener D, Zubke W. Laparoscopic supracervical hysterectomy using EnSeal vs standard bipolar coagulation technique: randomized controlled trial. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):661-6. doi: 10.1016/j.jmig.2013.04.014. Epub 2013 Jun 20. PMID 23791399
- [Derived] Rothmund R, Szyrach M, Reda A, Enderle MD, Neugebauer A, Taran FA, Brucker S, Hausch A, Wallwiener C, Kraemer B. A prospective, randomized clinical comparison between UltraCision and the novel sealing and cutting device BiCision in patients with laparoscopic supracervical hysterectomy. Surg Endosc. 2013 Oct;27(10):3852-9. doi: 10.1007/s00464-013-2994-4. Epub 2013 May 14. PMID 23670744